CLINICAL TRIAL: NCT02602899
Title: Deep Brain Stimulation of the Anterior Nucleus of the Thalamus in Refractory Epilepsy
Acronym: ANT-DBS-RE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-013
Record Dates: First submitted 2015-10-10; First posted 2015-11-11 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Refractory Epilepsy
Keywords: PINS; Deep Brain Stimulator; Refractory Epilepsy; Anterior Thalamic Nucleus
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PINS Deep Brain Stimulator (Experimental): Deep Brain Stimulator is on,continuous stimulation to the brain,
  Interventions: Procedure: PINS'Deep Brain Stimulator device

INTERVENTIONS:
Procedure: PINS'Deep Brain Stimulator device — deep brain stimulation of the PINS'IPG function to anterior nucleus of the thalamus is off in a short time

SUMMARY:
Evaluate the long-term clinical effectiveness and safety of the PINS Deep Brain Stimulation to patients with refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* age 12-60.
* having tried at least two appropriate anti-epileptic drugs (AEDs) tested to tolerance or to blood levels at upper end of the target range of which at least 2 have been tolerated at normal dose.
* at least 6 seizures per month.
* in good health except epilepsy.
* to with normal MMSE score
* patients or his(her) familys could understand this method and sign the informed consent 7）Patients with good compliance and could complete postoperative follow-up

Exclusion Criteria:

* results of MRI remind epilepsy caused by intracranial space-occupying lesions.
* the vagus nerve lesion and damage
* tumor, cardiopulmonary anomaly, progressive neurological diseases, asthma，mental disease，peptic ulcer，diabetes Type 1，bad health etc, and other surgical contraindication.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluation period 6 month | 6 month of stimulation

SECONDARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluation period | 1,3,6,12 months of stimulation
Overall Quality of Life in Epilepsy-31 (QOLIE-31) Score in Patients With Baseline & at Least One Post-baseline QOLIE Assessment | Mean change from baseline QOLIE-31 Overall Score at 1,3,6,12 months
Change in the Number of Anti-epileptic Drugs Prescribed | At 1,3,6,12 months
Change from Baseline in the Engel and McHugh description | At 1,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luming Li, Study Chair — study principal investigator
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China